CLINICAL TRIAL: NCT03577678
Title: Comminuted Lateral Half Fracture of Clavicle is Most Common and at This Case Report Study the Investigators Introduce a New Prophesies for This Fracture
Brief Title: New Prosthesis for Comminuted Fracture of Lateral Half of Clavicle
Acronym: Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sahar Ahmed Abdalbary, Principal investigator., Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Cairo University Hospital
Record Dates: First submitted 2018-06-13; First posted 2018-07-05 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Bone Fracture; Bone Lesion; Clavicle Fracture
Keywords: Comminuted lateral clavicle fracture , New prosthesis,
MeSH Terms: conditions — Fractures, Bone | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Surgery was made to fix the new prosthesis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- observational (Experimental): orthopaedic Surgery to fix lateral half prosthesis for clavicle
  Interventions: Procedure: Surgery to fix lateral half prosthesis for clavicle

INTERVENTIONS:
Procedure: Surgery to fix lateral half prosthesis for clavicle — Surgery to fix lateral half prosthesis for clavicle
  Other Names: surgery

SUMMARY:
This study to evaluate the efficacy of new prosthesis in treatment of comminuted fracture of lateral half of the clavicle in adult female.

DETAILED DESCRIPTION:
. Lateral clavicle fracture lead to sever pain and affect on shoulder movement . This prosthesis will compensate the lost part of the clavicle due to fracture to return the patient to the daily living activity without pain.

This prosthesis will reconstruct the missed part of the clavicle.

ELIGIBILITY:
Inclusion Criteria:

* Female has right lateral part comminuted fracture clavicle .

Exclusion Criteria:

* Male patient
* Cancer bone patient.
* Pregnant
* Left lateral part comminuted fracture clavicle

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-08-05 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
CT scan | 1 Day
  CT scan to determine the status and position of the prosthesis

SECONDARY OUTCOMES:
CT scan | 6 month
  CT scan to determine the status and position of the prosthesis
Pain intensity measurements: Visual analogue scale | 6 month
  Visual analogue scale from 0 to 10 , 0 is no pain and 10 unbearable pain
American shoulder and elbow surgeons score Special Score for shoulder pain and function. | 6 month
  The American shoulder and elbow surgeons score is a composite instrument, requiring both a physician assessment and a patient-completed portion.
  . This includes a section on pain (7 items) and a section on activities of daily living (10 items). Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
  Intensity of pain: 0; Putting on a coat is not difficult; Sleeping on the affected side is not difficult; Washing my back/doing up my bra is not difficult; Managing toiletting is not difficult; Combing my hair is not difficult; Reaching a high shelf is not difficult; Lifting 10lbs. (4.5kg) above my shoulder is not difficult; Throwing a ball overhand is not difficult; Doing my usual work is not difficult; Doing my usual sport/leisure activity is not difficult; It means good shoulder.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar A Abdalbary, ph.D., Principal Investigator
Locations (1):
- Alkasr alini hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No